CLINICAL TRIAL: NCT01299155
Title: A Randomized, Pilot Study, Subject Masked Comparison of Visual Function After Bilateral Implantation of Presbyopia Correcting Intraocular Lenses (IOLs)
Brief Title: A Comparison of Visual Function After Bilateral Implantation of Presbyopia Correcting Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M10-070
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2011-10

CONDITIONS: Cataract
Keywords: Intraocular Lens; Presbyopia Correcting IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReSTOR +3 (Experimental): Bilateral implantation of a ReSTOR +3 Intraocular Lens (IOL) Model SN6AD1
  Interventions: Device: ReSTOR +3
- LENTIS MPlus (Active Comparator): Bilateral implantation of a LENTIS MPlus Intraocular Lens (IOL) Model
  Interventions: Device: LENTIS MPlus

INTERVENTIONS:
Device: ReSTOR +3 — Bilateral implantation of an Alcon AcrySof ReSTOR +3 Intraocular Lens (IOL) Model SN6AD1 following cataract extraction.
  Arms: ReSTOR +3
Device: LENTIS MPlus — Bilateral implantation of a LENTIS MPlus Intraocular Lens (IOL) following cataract extraction.
  Arms: LENTIS MPlus

SUMMARY:
To prospectively evaluate postoperative visual and refractive parameters in a series of subjects bilaterally implanted with AcrySof ReSTOR +3 vs. those bilaterally implanted with LENTIS MPlus Intraocular Lens (IOL).

ELIGIBILITY:
Inclusion Criteria:

* are willing and able to understand and sign an informed consent
* <= 1.0 Diopters of regular corneal astigmatism in both eyes. NOTE: look for consistency between manual keratometry, auto-keratometry and simulated keratometry measures to ensure "regular" astigmatism prior to enrollment. Subjects who wear contact lenses must discontinue its use for at least 2 weeks (soft contact lens) and at least 3 weeks (gas permeable contact lens) and until corneal topography shows stability prior to preoperative study measurements.
* are willing and able to attend postoperative examinations per protocol schedule
* are more than 21 years of age, of either gender and any race:
* require bilateral cataract extraction followed by posterior intraocular lens (IOL) implantation used as on-label procedure
* be willing to have second eye surgery within one month of first eye surgery
* are in good ocular health, with the exception of cataracts
* are free of disease(s)/condition(s) listed in the "Precautions" section of the AcrySof IQ ReSTOR +3 and LENTIS Mplus package inserts
* are able to read and understand one of the following languages: Dutch or Spanish

Exclusion Criteria:

* Planned multiple procedures, including limbal relaxing incision (LRI), during cataract/IOL implantation surgery
* An ocular disease and/or condition that may compromise visual acuity levels (i.e. glaucoma, diabetic retinopathy, macular degeneration, amblyopia, pupil abnormality such as corectopia, etc.)
* Previous corneal surgery and/or reshaping
* Clinically significant corneal endothelial dystrophy (e.g. Fuchs' dystrophy)
* History of corneal disease (eg. herpes simplex, herpes zoster keratitis, etc.)
* History of retinal detachment
* Subjects that have an acute or chronic disease or illness that would increase the operative risk or confound the results of this investigation (eg, immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness).
* suturing of incision required at time of surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Unilateral Uncorrected Near Visual Acuity | 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Oviedo, Principality of Asturias, Spain